CLINICAL TRIAL: NCT01486459
Title: A Feasibility Trial Using Lithium As A Neuroprotective Agent In Patients Undergoing Prophylactic Cranial Irradiation For Small Cell Lung Cancer
Acronym: TULIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruits
Sponsor: Barwon Health (Other Government)
Collaborators: Deakin University (Other); Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALCC 11.01
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2013-08

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCI with lithium (Experimental): Prophylactic cranial irradiation Lithicarb® tablets 250mg/day for 6 weeks. Initial dosing will be 250mg given once daily, and increased by 250 - 500 mg increments depending on plasma levels.
  Interventions: Drug: Lithium
- Standard (No Intervention): Prophylactic cranial irradiation alone.

INTERVENTIONS:
Drug: Lithium — 250 mg daily for 6 weeks, increased 250 - 500 mg depending on plasma levels.
  Other Names: Lithicarb
  Arms: PCI with lithium

SUMMARY:
Small cell lung cancer is an aggressive neuroendocrine tumour that often presents with extensive (metastatic) disease. Chemotherapy is the mainstay of treatment, with radiotherapy to the primary tumour. It is now part of care to also offer Prophylactic Cranial Irradiation (PCI) in order to prevent spread of the cancer into the brain.

Cognitive impairment can result after cranial irradiation. Lithium is thought to be neuroprotective. It is hypothesized that lithium administration with PCI will be safe, tolerable and feasible, and can be studied to prevent or ameliorate the ensuing cognitive impairment.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is an aggressive neuroendocrine tumour that often presents with extensive (metastatic) disease.[1] It frequently has micrometastatic disease at presentation. Chemotherapy is the mainstay of treatment with radiotherapy to the primary tumour. It is now part of care to offer Prophylactic Cranial Irradiation (PCI)with 25 Gy in 10 fractions dependent on the extent of response in the primary tumour and the patient's performance status. PCI is routine care for limited stage patients showing response and can be considered in selected patients with limited stage disease showing good response.Somnolence syndrome is a common intermediate side effect of cranial radiotherapy that occurs about six weeks after treatment and manifests as lethargy, increased sleepiness and poor attention or subtle memory changes and altered temperament[2].

The use of cranial irradiation is linked to neurocognitive complications such as long term memory, mood and concentration issues[3]. Decline in attention, executive function, motor, language and general intellectual skills have all been reported. There is the suggestion of a more rapid progression of dementing illness in patients receiving cranial irradiation although the numbers of long term survivors is limited[3]. Radiation mediates neurocognitive effects by affecting glial cells, neural stem and progenitor cells[4, 5] and the vascular structures[3, 6]. Cranial irradiation delivered to mice has been shown to reduce neural proliferation translating to long term reduction in neurogenesis[7, 8]. Lithium confers neuroprotection and is associated with less cognitive loss in various brain injury models including after cranial irradiation[9, 10]. In addition, neural stem/progenitor cells positively respond to Lithium treatment under basal conditions[11, 12]. In humans, 4 weeks of Lithium increases brain grey matter content[13] and hippocampal volume[14] as evidenced by MRI scanning. Lithium was found to protect irradiated hippocampal neurons in mice from apoptosis resulting in better performance reflecting learning and memory function[10]. Lithium is known to reduce oxidative stress, specifically via the glutathione system. Lithium is a standard part of the management of moderate to severe bipolar disorder and schizoaffective disorders and its toxicity profile is well understood[15, 16]. In bipolar disorder, lithium has been shown to prevent the loss of cortical grey matter that occurs as part of the neuroprogressive cascade seen in the disorder[17]. There is limited prospective clinical data regarding the use of lithium as a neuroprotectant. A large Danish observational cohort study, demonstrated that use of lithium (in those with mood disorders, who display an increased risk for dementia) was associated with reduction of the rate of dementia to the same level as that for the general population[18]. A follow up study by the same group showed similar findings[19]. A metaanalysis of lithium on cognitive performance demonstrated minor negative effects on cognition[20]. There has been one early phase study using lithium as a neuroprotective agent presented in abstract form at the 2007 American Society for Therapeutic Radiology and Oncology (ASTRO)[21] and updated at the 2008 annual meeting of the Society of NeuroOncology (SNO)[22].

Long term lithium treatment has also shown promise in amnestic mild cognitive impairment in a study that randomized 45 participants to receive lithium (0.25-0.5 mmol/l) (n = 24) or placebo (n = 21) in a 12 month, doubleblind trial[23]. Lithium treatment was associated with a significant decrease in CSF concentrations of Ptau(P =0.03) and better performance on the cognitive subscale of the Alzheimer's Disease Assessment Scale and in attention tasks. The data support the notion that lithium has disease modifying properties with potential clinical implications in the prevention of Alzheimer's disease.[23]

References:

1. Turrisi AT, 3rd, Kim K, Blum R et al. Twice daily compared with once daily thoracic radiotherapy in limited small cell lung cancer treated concurrently with cisplatin and etoposide. N England J Med 1999; 340: 265271.
2. Kelsey CR, Marks LB. Somnolence syndrome after focal radiation therapy to the pineal region: case report and review of the literature. J Neurooncol 2006; 78: 153156.
3. Armstrong CL, Gyato K, Awadalla AW et al. A critical review of the clinical effects of therapeutic irradiation damage to the brain: the roots of controversy. Neurophysiol Rev 2004; 14: 6586.
4. Monje ML, Vogel H, Masek M et al. Impaired human hippocampal neurogenesis after treatment for central nevrous system malignancies. Ann Neurol. 2007; 62, 515520.
5. Monje ML, Palmer T. Radiation injury and neurogenesis. Curr Opin Neurol. 2003; 129134.
6. Perry A, Schmidt RE. Cancer therapy associated CNS neuropathology: an update and review of the literature. Acta Neuropathol 2006; 111: 197212.
7. Rola R, Raber J, Rizk A et al. Radiation induced impairment of hippocampal neurogenesis is associated with cognitive deficits in young mice. Exp Neurol 2004; 188: 316330.
8. Vorhees CV, Williams MT. Morris water maze procedures for assessing spatial and related forms of learning and memory. Nat Protoc 2006; 1: 848858.
9. Rowe MK, Chuang DM. Lithium neuroprotection: molecular mechanisms and clinical implications. Expert Rev Mol. Med. 2004;6: 118.
10. Yazlovitskaya EM, Edwards E, Thotala D et al. Lithium treatment prevents neurocognitive deficit resulting from cranial irradiation. Cancer Res 2006; 66: 1117911186.
11. Chen G, Rajokowska G, Du F et al. Enhancement of hippocampal neurogenesis by lithium. J. Neurochem. 2000; 75: 17291734.
12. Yan XB, Hou HL, Wu LM et al. Lithium regulates hippocampal neurogenesis by ERK pathway and facilitates recovery of spatial learning and memory in rats after transient global cerebral ischemia. Neuropharmacology 2007;53: 487495.
13. Moore GJ, Bebchuk JM, WIlds IB et al. Lithium induced increase in human brain grey matter. Lancet 2000; 356:12411242.
14. Foland LC, Altshuler LL, Sugar CA et al. Increased volume of the amygdala and hippocampus in bipolar patients treated with lithium. Neuroreport 2008;19:221224.
15. Dowdan J. Therapeutic Guidelines: Psychotropic. (Version 5). Melbourne: 2003.
16. Foutoulakis KN, Vieta E, SanchezMoreno J et al. Treatment guidelines for bipolar disorder: a critical review. J Affect Disord 2005; 86:110.
17. Berk M, Kapczinski F, Andreazza AC et al. Pathways underlying neuroprogression in bipolar disorder: focus on inflammation, oxidative stress and neurotrophic factors. Neurosci Biobehav Rev 2011; 35:804817.
18. Kessing LV, SOndergard L, Forman JL, Andersen PK. Lithium treatment and risk of dimential. Arch Gen Psychiatry 2008; 65: 13311335.
19. Kessing LV, Forman JL, Andersen PK. Does lithium protect against dementia? Bipolar Disord 2010; 12: 8794.
20. Wingo AP, Wingo TS, Harvey PD, Baldessarini RJ. Effects of lithium on cognitive performance: a metaanalysis. J. Clin Psychiatry 2009; 70: 15881597.
21. Yang ES, Lu B, Hallahan DE. Lithium mediated neuroprotection during cranial irradiation: A phase 1 trial. In ASTRO (American SOciety for Therapeutic Radiology and Oncology) 49th Annual Conference. Los Angeles CA:

2007 [22] Xia F, Yang E, Hallahan D, Lu B. Lithium mediated neuroprotection during cranial irradiation: a phase I trial. Neurooncology 2008; 10: 887887.

[23] Forlenza OV, Diniz BS, Radanovic M et al. Disease modifying properties of long term lithium treatment for amnestic mild cognitive impairment: randomized controlled trial. The British Journal of Psychiatry: The Journal of Mental Science 2011; 198: 351356.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed high grade small cell neuroendocrine carcinoma.
* Patients can either have:

  * Limited stage disease with CR or PR OR
  * Extensive stage disease with CR or good PR
* Patients must have discontinued other chemotherapies at least 3 weeks prior to randomisation.
* Prior radiation therapy to the chest is allowed but must be completed at least 3 weeks prior to randomisation.
* ECOG Performance Status 0 to 2.
* Adequate bone marrow, liver, and renal function as assessed by the following:

  * Hemoglobin ≥ 9.0 g/dl
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Total bilirubin ≤ 2.0 times the upper limit of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (≤ 5x ULN for patients with liver involvement)
  * International Normalized Ratio for Prothrombin Time (PT-INR) ≤ 1.5 and activated partial prothrombin time (aPTT) within 5% of normal limits for patient NOT on anticoagulation.
  * Estimated Glomerular Filtration Rate (eGRF) > 50 ml/min .
* Male or female aged >18 years
* Patients must be able and willing to sign a written informed consent. A signed informed consent must be appropriately obtained prior to any study specific procedures.
* Patients must be able to swallow and retain oral medication.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to randomisation and must agree to use adequate contraception prior to randomisation and for the duration of study participation.

Exclusion Criteria:

* Life expectancy less than 3 months.
* Substance abuse, medical, psychological, or social condition that may interfere with the patient's participation in the study or evaluation of the study results.
* Severe cardiac or renal disease.
* Frank hypothyroidism.
* Hyponatraemia.
* Known or suspected allergy to lithium.
* Women who are pregnant or breast-feeding.
* Inability to comply with protocol and /or not willing or not available for follow-up assessments.
* Significant psychiatric or neurologic illness (prior known psych/cognitive/CNS pathology eg CVA; known or prior brain metastases
* Current lithium therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of a project design where the patients are randomized into lithium or placebo | 1 year
  Number of participants with adverse events

SECONDARY OUTCOMES:
Neurocognition | 1 year
  Measurements of CogState, Cognitive Failures Questionnaire, CES-D and somnolence syndrome using the Epworth Sleepiness Scale in patients treated with lithium compared to the controls

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MD, Principal Investigator — Barwon Health
Locations (2):
- Australia (2):
  - Barwon Health, Geelong, Victoria
  - Peter MacCallum Cancer Centre, Moorabbin, Victoria